CLINICAL TRIAL: NCT01583816
Title: Prospective, Randomized, Partly Blinded, in Part Placebo-controlled, Multicenter, Dose-finding Trial Exploring Safety, Tolerability and Efficacy of a Topical Resiquimod Gel in Patients With Multiple Actinic Keratosis Lesions
Brief Title: Dose-finding, Safety, Efficacy Trial of Topical Resiquimod in Patients With Multiple Actinic Keratosis Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP848-AK-1101
Record Dates: First submitted 2012-04-18; First posted 2012-04-24 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Resiquimod
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Resiquimod Gel 0.03% or placebo (Experimental): Resiquimod gel 0.03% or placebo, once daily, 3x per week for 4 weeks, break of 8 weeks, repeated once
  Interventions: Drug: Resiquimod 0.03%; Drug: placebo
- Resiquimod or placebo (Experimental): Once daily, 7x within 2 weeks, break of 8 weeks, cycle repeated once
  Interventions: Drug: Resiquimod 0.03%; Drug: placebo
- Resiquimod or vehicle (Experimental): Once daily, 5x for 1 week, break of 8 weeks, cycle repeated once
  Interventions: Drug: Resiquimod 0.03%; Drug: placebo
- Resiquimod gel 0.01% (Experimental): Once daily, 3x/week until occurrence of biological endpoint or for a maximum of 8 weeks (no repetition of cycle), 8 weeks follow-up
  Interventions: Drug: Resiquimod 0.01%
- Resiquimod gel 0.03% (Experimental): Once daily, 3x/week until occurrence of biological endpoint or for a maximum of 8 weeks (no repetition of cycle), 8 weeks follow-up
  Interventions: Drug: Resiquimod 0.03%

INTERVENTIONS:
Drug: Resiquimod 0.03% — topical application
  Arms: Resiquimod Gel 0.03% or placebo; Resiquimod gel 0.03%; Resiquimod or placebo; Resiquimod or vehicle
Drug: Resiquimod 0.01% — topical application
  Arms: Resiquimod gel 0.01%
Drug: placebo — topical application
  Arms: Resiquimod Gel 0.03% or placebo; Resiquimod or placebo; Resiquimod or vehicle

SUMMARY:
A Dose-Finding Study of Resiquimod Evaluating Safety and Efficacy in Patients with Multiple Actinic Keratosis Lesions

DETAILED DESCRIPTION:
Prospective, randomized, partly blinded, in part placebo-controlled, multicenter dose-finding trial with patients suffering from AK. Patients were observed for efficacy, local tolerability and safety. A total of 14 sites in Switzerland and Germany enrolled male and female patients over 18 years of age with clinically diagnosed AK lesions Patients were randomized to receive resiquimod gel (Treatment Arms 1, 2, 3, 4, or 5) or matching vehicle (Treatment Arms 1-Pla, 2-Pla, or 3-Pla):

Treatment Arms 1, 2 and 3: The patient was randomly assigned to one of three treatment groups and within each group there was one randomly assigned placebo patient for every two treatment patients (parallel-group randomization; 2:1 active vs placebo).

Treatment Arms 4 and 5: The patient was randomly assigned to one of two treatment groups (parallel-group randomization, 1:1).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or nonpregnant, nonlactating female, ≥18 years
* A minimum of 2 clinically diagnosed AK-lesions within a defined area (25 cm2 contiguous treatment area). One AK-lesion must have a diameter of at least 6 mm (indicator lesion)
* AK-lesions on balding scalp, forehead or face

Exclusion Criteria:

* Known allergy or hypersensitivity to any of the trial gel ingredients
* Dermatological disease or condition that might be exacerbated by resiquimod gel treatment or may impair trial assessments
* Evidence of unstable or uncontrolled clinically significant medical conditions, active infection, immunosuppression or systemic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete clinical clearance in the treated area at the end of trial | 8 weeks after a maximal treatment period of 8 weeks

SECONDARY OUTCOMES:
Evaluation of adverse events (AEs) and serious adverse events (SAEs) | up to 24 weeks
Evaluation of local tolerability (burning, itching, sensation of pain) by means of symptom scoring scales | up to 24 weeks
Number of patients with partial clearance | 8 weeks after a maximal treatment period of 8 weeks
Evaluation of systemic tolerability [hematology, blood chemistry, vital signs] | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars E French, MD, Principal Investigator — University Clinic of Dermatology, Zurich
Locations (10):
- Germany (5):
  - Hauttumorcentrum Charité (HTCC), Berlin
  - Medizinisches Zentrum Bonn - Friedensplatz, Bonn
  - Hautzentrum, Düsseldorf
  - Johannes Wesling Klinikum Minden, Minden
  - KLINIKUM VEST GmbH Knappschaftskrankenhaus, Recklinghausen
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitaetsspital Zurich, Zurich